CLINICAL TRIAL: NCT05499182
Title: Identification of Implementation Strategies to Promote Depression Treatment Use Among Latino Adolescents
Brief Title: Latino Teen Depression Treatment Study
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00110026
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Depression
Keywords: Adolescent; Latino; Depression; Treatment
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Teens: Teens are: 1) Male 2) Aged 13-17; 3) self-identified as Hispanic/Latino; 4) diagnosed with Major Depressive Disorder or Persistent Depressive Disorder/Dysthymia; and 5) referred to psychotherapy or prescribed medication for depression. Teens will be excluded if they are experiencing intense psychological distress or imminent thoughts of suicide.
- Parents: Parents will 1) Be parents or legal guardians of teens; and 2) Speak and read English or Spanish.
- Healthcare Providers: Healthcare providers will 1) Self-identify as regularly providing clinical care to Latino adolescents with depression; and 2) be in a role in which they can refer to or provide depression treatment.

SUMMARY:
Despite experiencing higher rates of depressive symptoms (Center for Disease Control and Prevention, 2020) and similar rates of Major Depressive Disorder (MDD; Substance Abuse and Mental Health Services Administration (SAMHSA), 2019), Latino adolescents in the U.S. are significantly less likely than their non-Latino White peers to receive treatment for MDD (SAMHSA, 2019). The purpose of this study is to identify a stakeholder-preferred implementation strategy that may improve psychotherapy attendance among Latino adolescents. Latino adolescent-parent dyads and healthcare providers will be recruited from healthcare settings and social media. Focus groups will be conducted with healthcare providers (n=5), and individual interviews will be conducted with Latino adolescents with a diagnosis of depression (n=15) and their parents (n=15).

ELIGIBILITY:
Inclusion Criteria for Teens:

* Male gender
* Aged 13-17 years
* Diagnosed with Major Depressive Disorder or Persistent Depressive Disorder
* Referred to psychotherapy and/or prescribed antidepressant medications for depression

Exclusion Criteria for Teens:

* Experiencing imminent thoughts of self-harm or suicide
* Experiencing acute psychological distress (e.g., uncontrolled crying)

Inclusion Criteria for Parents:

* Parent or legal guardian of teen
* Able to read and speak English or Spanish

Exclusion Criteria for Parents:

* Unable to read/speak English or Spanish

Inclusion Criteria for Healthcare Providers:

* Self-identification as regularly providing clinical care to Latino adolescents with depression
* Be in a role in which they can provide or refer patients to depression treatment

Exclusion Criteria for Healthcare Providers

* Unable to provide or refer to depression treatment

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Teens will be required to self-report a male gender. Parent and healthcare provider participants will not be recruited according to gender.
Study Population: Three samples will be recruited on a national scale: Latino male teens diagnosed with depression, their parents/guardians, and healthcare providers (behavioral health and primary care) who regularly care for Latino adolescents.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Preferred implementation strategy to improve depression treatment use generated from qualitative interviews/focus groups | Baseline
  Implementation strategy preference options will include: 1) Near Peer Depression Support Groups; 2) Parent-Teen Depression Treatment Activation Training; and 3) Depression Care Navigation Services. We will determine which strategy is most preferred by asking stakeholders, "Which of these strategies would work best for you/your family/Latino teens?" We will add up the responses to determine the preferred strategy with the highest frequency.

SECONDARY OUTCOMES:
Number of barriers to depression treatment use generated from qualitative interviews/focus groups | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Allison M Stafford, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Researchmatch.org, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Due to the qualitative nature of this study, we will not be sharing participant data with other researchers.